CLINICAL TRIAL: NCT01026090
Title: A Phase IV, Double-blind, Placebo-controlled, Canadian Multicentre Study Comparing Two Treatment Strategies of Dronedarone Administration Following ELECTive caRdioversion for Prevention of Symptomatic Atrial Fibrillation (AF) Recurrence
Brief Title: Dronedarone Pattern of Use in Patients Scheduled for Elective Cardioversion (ELECTRA)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: 'Sponsor decision following recruitment issues, not related to any safety concerns in the study
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRONE_L_04742
Record Dates: First submitted 2009-12-02; First posted 2009-12-04 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dronedarone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dronedarone pre-cardioversion (Experimental): Dronedarone 400 mg twice a day for 5-7 days prior to cardioversion, then dronedarone 400 mg twice a day for 6 months after cardioversion
  Interventions: Drug: Dronedarone
- Placebo pre-cardioversion (Placebo Comparator): Placebo (for dronedarone) twice a day for 5-7 days prior to cardioversion, then dronedarone 400 mg twice a day for 6 months after cardioversion
  Interventions: Drug: Dronedarone; Drug: Placebo (for dronedarone)

INTERVENTIONS:
Drug: Dronedarone — Film-coated tablet
  Oral administration under fed conditions (during breakfast and dinner)
  Other Names: MULTAQ; SR33589
Drug: Placebo (for dronedarone) — film-coated tablet strictly identical in appearance
  Oral administration under fed conditions (during breakfast and dinner)
  Arms: Placebo pre-cardioversion

SUMMARY:
Primary Objective:

To determine whether daily administration of dronedarone started 5-7 days before cardioversion is superior to dronedarone started only after cardioversion with respect to the absence of symptomatic, ECG confirmed, atrial fibrillation (AF) recurrence over 6 months in adult patients with persistent AF, for whom cardioversion is clinically indicated and planned to reduce symptoms and antiarrhythmic treatment is clinically indicated to reduce the risk of cardiovascular hospitalization due to AF.

Secondary Objectives:

Main Secondary :

* To assess the number of symptomatic AF recurrences/patient/6 months with and without ECG confirmation;
* To assess characteristics of symptomatic AF recurrence in the two treatment arms (frequency, duration of episodes, type, number, and severity of AF symptoms per patient);
* To compare the rates of early recurrences of AF between the two treatment strategies;

Other secondary:

* To assess whether there is a difference in proportion of patients with symptomatic AF recurrences (with and without ECG confirmation) between the two treatment strategies;
* To assess whether there is a difference in number of electrical cardioversions per patient between the two treatment strategies;
* To assess the impact of the two strategies on number of shocks, cumulative amount of energy delivered, shock failure, and immediate success of cardioversion;
* To assess whether there is a difference in rate of cardiovascular (CV) hospitalizations and length of hospital stay between the two treatment strategies;
* To assess whether there is a difference in quality of life between the two treatment strategies.

DETAILED DESCRIPTION:
The study period of approximatively 6 months consisted in:

* Double-blind treatment period (placebo or dronedarone) for 5-7 days prior to cardioversion;
* Electrical cardioversion;
* Open-label treatment period with dronedarone for 6 months after cardioversion.

ELIGIBILITY:
Inclusion criteria:

- Adult patients with persistent AF (current episode at the screening visit >72 hrs and <12 month duration), for whom cardioversion was clinically indicated and planned to reduce symptoms and antiarrhythmic treatment was clinically indicated to reduce the risk of cardiovascular hospitalization due to AF.

Exclusion criteria:

* Severe congestive heart failure (NYHA Class IV) and other unstable hemodynamic conditions;
* Bradycardia <50 bpm;
* QTc Bazett interval ≥500 ms;
* Second- or third- degree atrio-ventricular (AV) block, or sick sinus syndrome (except when used in conjunction with a functioning pacemaker);
* Severe hepatic impairment;
* Pregnancy and lactation;
* History of hypersensitivity reactions to dronedarone or any of its excipients or component of the container.

Concomitant drugs:

* Antiarrhythmic drugs (AADs) other than dronedarone should not be administered during the study and should be withdrawn for at least five plasma half-lives prior to the first study drug administration;
* Dronedarone should not be co-administered with strong CYP3A4 inhibitors;
* Dronedarone should not be co-administered with drugs inducing torsades de pointes.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2009-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with at least one symptomatic, ECG confirmed, AF recurrence | 6 months from initial cardioversion

SECONDARY OUTCOMES:
Number of Symptomatic AF Recurrences/Patient/6 Months (With or Without ECG Confirmation) | up to 6 months from initial cardioversion
Characteristics of Symptomatic AF Recurrence (Frequency, Duration of Episodes, Type, Number, and Severity of AF Symptoms) | up to 6 months from initial cardioversion
Proportion of Participants With Early Recurrence of AF (i.e. From 5 Minutes to to 7 Days Following Cardioversion) | up to 7 days following initial cardioversion
Proportion of Participants With Symptomatic AF Recurrences (With or Without ECG Confirmation) | up to 6 months from initial cardioversion
Number of Electrical Cardioversions Per Patient | up to 6 months from intial cardioversion
Number of Shocks Required During Initial Cardioversion | during the initial cardioversion
Cumulative Amount of Energy Delivered and Shock Failure | during the initial cardioversion
Proportion of Participants With Immediate Recurrence of AF (From 5 Seconds to 5 Minutes After Electrical Shock) | during the initial cardioversion
Number of CV Hospitalizations | up to 6 months from initial cardioversion
Quality of Life, as Measured by Atrial Fibrillation Severity Scale (AFSS) and Atrial Fibrillation Effect on Quality of Life (AFEQT) Questionnaires | Baseline and 6 months after initial cardioversion

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (43):
- Canada (43):
  - Investigational Site Number 1240033, Abbotsford
  - Investigational Site Number 1240026, Barrie
  - Investigational Site Number 1240050, Calgary
  - Investigational Site Number 1240010, Cambridge
  - Investigational Site Number 1240049, Edmonton
  - Investigational Site Number 1240005, Granby
  - Investigational Site Number 1240021, Greater Sudbury
  - Investigational Site Number 1240039, Greater Sudbury
  - Investigational Site Number 1240001, Greenfield Park
  - Investigational Site Number 1240046, Grimsby
  - Investigational Site Number 1240040, Hamilton
  - Investigational Site Number 1240037, Hamilton
  - Investigational Site Number 1240044, Kingston
  - Investigational Site Number 1240029, Kitchener
  - Investigational Site Number 1240013, Laval
  - Investigational Site Number 1240043, Lévis
  - Investigational Site Number 1240038, Maple Ridge
  - Investigational Site Number 1240023, Montreal
  - Investigational Site Number 1240006, Montreal
  - Investigational Site Number 1240008, Montreal
  - Investigational Site Number 1240018, Newmarket
  - Investigational Site Number 1240012, Niagara Falls
  - Investigational Site Number 1240020, North York
  - Investigational Site Number 1240015, Oshawa
  - Investigational Site Number 1240036, Oshawa
  - Investigational Site Number 1240024, Ottawa
  - Investigational Site Number 1240032, Ottawa
  - Investigational Site Number 1240056, Red Deer
  - Investigational Site Number 1240003, Saint-Charles-Borromée
  - Investigational Site Number 1240053, Saskatoon
  - Investigational Site Number 1240016, Scarborough
  - Investigational Site Number 1240027, Sherbrooke
  - Investigational Site Number 1240007, St. Georges
  - Investigational Site Number 1240041, St. John's
  - Investigational Site Number 1240002, Ste-Foy
  - Investigational Site Number 1240025, Toronto
  - Investigational Site Number 1240011, Toronto
  - Investigational Site Number 1240019, Toronto
  - Investigational Site Number 1240009, Trois-Rivières
  - Investigational Site Number 1240047, Vancouver
  - Investigational Site Number 1240035, Victoria
  - Investigational Site Number 1240014, Willowdale
  - Investigational Site Number 1240051, Windsor